CLINICAL TRIAL: NCT00733109
Title: Management of Cervical Intraepithelial Neoplasia Grade 2
Acronym: CIN2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Jose Lucio Martins Machado, UNICID- School of Medical Sciense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIN 2
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2008-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: CIN2; management
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- excision of the lesion (Active Comparator)
  Interventions: Procedure: Excision of the lesion
- espontaneous regression (No Intervention)
  Interventions: Other: Follow-up for spontaneous regression of the lesion

INTERVENTIONS:
Procedure: Excision of the lesion — Surgery with Large Loop Excision of Transformation Zone (LLETZ)
  Other Names: LEETZ
  Arms: excision of the lesion
Other: Follow-up for spontaneous regression of the lesion — Follow-up at last 12 months
  Other Names: conservative managment
  Arms: espontaneous regression

SUMMARY:
The aim of this study was to compare two management options for CIN 2. This randomized clinical trial performed between 2003 and 2006. A series of 90 Brazilian women diagnosed as CIN2 were randomized into two groups: 1) 45 whose lesion was excised and,2) 45 women subjected to follow-up at 3-month intervals for 12 months.

DETAILED DESCRIPTION:
Pap smear and colposcopy were performed at every follow-up visit and all lesions were completely visible at colposcopy.

The researchers purpose was to make some comments about the over treatment and the misclassification of CIN 2.

ELIGIBILITY:
Inclusion Criteria:

* Histological CIN2 diagnosis

Exclusion Criteria:

* Previous CIN treatment

Ages: 18 Years to 61 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2003-03; Primary Completion 2006-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
43 women in the follow-up group, 44.1% experienced spontaneous regression, 20.9% had partial regression, 23.2% progressed to CIN3, and 11.6% showed persistence. 44 women whose lesion was excised, the regression rate was 90.9% | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia F Brenna, MD, PhD, Principal Investigator — Universidade Cidade de Sao Paulo; Ana C Guedes, MD, PhD, Principal Investigator — Universidade Cidade de Sao Paulo; Kari J Sirjanen, MD, PhD, Study Chair — University of Turku; Luis C Zeferino, MD, PhD, Study Director — University of Campinas, Brazil
Locations (1):
- Leonor Mendes de Barros Maternity Hospital, São Paulo, São Paulo, Brazil